CLINICAL TRIAL: NCT03423550
Title: Development of a Rapid and Accurate Diagnostic Assay for Tuberculosis by Using New Sample Preparation and Detection Technique
Brief Title: Development of a Rapid and Accurate Diagnostic Assay for Tuberculosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sei Won Lee, Principal Investigator, Asan Medical Center
Other Study IDs: 2018-0020
Record Dates: First submitted 2018-01-28; First posted 2018-02-06 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants who are suspected with TB

SUMMARY:
This study evaluates new technique for diagnosis of tuberculosis. Among patients who are suspected with tuberculosis, participants will be tested conventional method including Xpert TB/RIF assay, and new diagnostic technique using homobifunctionalImidoesters compounds.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are suspected with pulmonary tuberculosis, tuberculosis meningitis, tuberculosis peritonitis, tuberculosis pleurisy

Exclusion Criteria:

* Under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients who are clinically suspected with pulmonary tuberculosis, tuberculosis meningitis, tuberculosis peritonitis, tuberculosis pleurisy
  * The participants will undertake conventional examination including AFB culture / smear and X-pert TB assay and new assay
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-01-16 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
The effectiveness of new diagnostic technique | An average of 2 year
  sensitivity and specificity of new test

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pulmonary and Critical Care Medicine and Clinical Research Center for Chronic Obstructive Airway Diseases, Asan Medical Center, University of Ulsan College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided